CLINICAL TRIAL: NCT07337655
Title: A Phase II/III Clinical Trial Evaluating the Efficacy and Safety of Aspirin and Lansoprazole in High-Risk Pregnant Women for the Prevention of Preterm Birth: A Biomarker-Enriched Design
Brief Title: Efficacy and Safety of Aspirin and Lansoprazole for Prevention of Preterm Birth in High-Risk Pregnant Women: A Biomarker-Enriched Trial
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Brice Gaudilliere, Professor of Anesthesiology, Perioperative and Pain Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 84662
Record Dates: First submitted 2026-01-09; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Pre-term Birth
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combination Therapy (Aspirin & Lansoprazole) (Experimental): Aspirin & Lansoprazole is taken once daily in the evening, preferably 30-60 minutes after dinner.
  Interventions: Drug: Low-Dose Aspirin Dose: 81 mg & Lansoprazole Dose: 30 mg
- Standard of Care (Other): Standard of Care
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Low-Dose Aspirin Dose: 81 mg & Lansoprazole Dose: 30 mg — 1. Low-Dose Aspirin Dose: 81 mg Route: Oral Frequency: Once daily Timing: Preferably in the evening; may be taken with food Duration: From randomization (12+0 to 16+6 weeks' gestation) until delivery
     Rationale:
     Low-dose aspirin has anti-inflammatory, antiplatelet, and placental perfusion-enhancing properties and is widely used in pregnancy for prevention of hypertensive disorders.
  2. Lansoprazole Dose: 30 mg Route: Oral Frequency: Once daily Timing: Preferably in the evening; may be taken with food Duration: From randomization (12+0 to 16+6 weeks' gestation) until delivery
  Rationale:
  Lansoprazole is a proton pump inhibitor with an established maternal-fetal safety profile. In addition to gastroprotection during aspirin therapy, it has immunomodulatory and anti-inflammatory effects that may act synergistically with aspirin to reduce pathways implicated in spontaneous preterm birth.
  Arms: Combination Therapy (Aspirin & Lansoprazole)
Other: Standard of Care — Standard of Care
  Arms: Standard of Care

SUMMARY:
This protocol describes a seamless Phase II/III, randomized, double-blind clinical trial evaluating the efficacy and safety of daily low-dose aspirin (81 mg) plus lansoprazole (30 mg) in pregnant individuals at high risk for preterm birth when compared to existing standard of care, identified through biomarker-enriched screening. Participants will be enrolled between 12-16+6 weeks' gestation and followed through delivery and postpartum. The primary objective is to determine whether the investigational combination reduces the incidence of preterm birth before 37 weeks of gestation compared with placebo.

DETAILED DESCRIPTION:
This study is a seamless Phase II/III, randomized, double-blind, biomarker-enriched clinical trial designed to evaluate the efficacy and safety of low-dose aspirin (81 mg daily) combined with lansoprazole (30 mg daily) for the prevention of preterm birth in pregnant individuals at high risk for spontaneous preterm delivery. Participants are enrolled early in pregnancy, between 12+0 and 16+6 weeks' gestation, and followed through delivery and a 6-week postpartum period.

Preterm birth remains a leading cause of neonatal morbidity and mortality, yet effective pharmacologic prevention strategies are limited, particularly following the withdrawal of 17-hydroxyprogesterone caproate. This trial addresses a critical unmet need by testing a repurposed, scalable, and globally accessible drug combination, guided by precision-medicine risk stratification rather than broad, unselected treatment.

Eligible participants are pregnant individuals aged 18 to 45 years with a singleton gestation who meet clinical high-risk criteria for preterm birth, such as a history of prior spontaneous preterm birth, cervical insufficiency, or short cervical length. All consented participants undergo biomarker screening, including a validated serum protein serological signature and/or a digital-twin immune profiling approach, to identify those at highest biological risk. Only participants who test biomarker-positive are eligible for randomization, ensuring an enriched population most likely to benefit from intervention.

Approximately 670 biomarker-positive participants will be randomized in a 1:1 ratio to one of two study arms: (1) daily aspirin plus lansoprazole in addition to standard obstetric care, or (2) standard obstetric care alone. Investigational therapy begins immediately after randomization and continues until delivery unless discontinued for safety or clinical indications. Standard obstetric care may include cervical length surveillance, vaginal progesterone, cerclage, and other guideline-based interventions, but excludes routine aspirin or proton pump inhibitor use unless clinically required outside the protocol.

The primary endpoint is the incidence of preterm birth before 37 weeks' gestation. Key secondary endpoints include preterm birth before 34 weeks, gestational age at delivery, hypertensive disorders of pregnancy, fetal growth restriction, neonatal morbidity, NICU admission, and perinatal mortality. Safety outcomes focus on maternal bleeding, gastrointestinal events, laboratory abnormalities, and serious maternal or neonatal adverse events. The study also evaluates treatment-biomarker interactions, longitudinal changes in immune and protein signatures, and concordance between predicted and observed treatment response.

The trial incorporates a group-sequential design with a pre-specified interim analysis during the Phase II portion to evaluate safety, biomarker performance, and conditional power, enabling a seamless transition to Phase III if criteria are met. Randomization is stratified by study site, prior preterm birth history, and biomarker category. Bias is minimized through centralized randomization, double blinding, standardized outcome definitions, intention-to-treat analysis, and oversight by an independent Data and Safety Monitoring Board (DSMB).

Conducted across multiple academic medical centers with expertise in maternal-fetal medicine, this study is designed not only to determine whether aspirin plus lansoprazole can reduce preterm birth, but also to generate high-quality evidence supporting a precision-guided preventive strategy. If successful, the trial has the potential to redefine pharmacologic prevention of preterm birth using safe, inexpensive, and widely available medications tailored to biologic risk.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 45 years at the time of informed consent.
* Pregnancy: Singleton intrauterine pregnancy confirmed by ultrasound.
* Gestational Age: Between 12+0 and 16+6 weeks' gestation at randomization, based on first- or early second-trimester ultrasound dating.
* Risk Status: At increased risk for spontaneous preterm birth, defined by at least one of the following:
* Prior spontaneous preterm birth (<37 weeks),
* History of second-trimester pregnancy loss related to cervical insufficiency,
* Short cervical length (≤25 mm) identified per site standard prior to randomization,
* Other clinically significant risk factors for spontaneous preterm birth as determined by the investigator.
* Biomarker Enrichment: Positive preterm birth risk classification based on serum protein signature and/or digital-twin immunologic profile, as defined in the protocol.
* General Health: In otherwise stable health, with medical conditions related to pregnancy risk permitted if well controlled.
* Informed Consent: Ability and willingness to provide written informed consent and comply with study procedures.
* Access to Care: Willingness to receive routine obstetric care at a participating study site and comply with follow-up through delivery and postpartum.

Exclusion Criteria:

1. Hypersensitivity / Contraindications

   * Known hypersensitivity, allergy, or intolerance to aspirin, other salicylates, lansoprazole, or other proton pump inhibitors (PPIs).
   * History of aspirin-exacerbated respiratory disease (AERD), including asthma, nasal polyps, or bronchospasm triggered by aspirin or other NSAIDs.
   * History of anaphylaxis or severe hypersensitivity to any component of the study drugs.
2. Hematologic / Bleeding Risk

   * History of major gastrointestinal bleeding, peptic ulcer hemorrhage, intracranial hemorrhage, or other serious bleeding disorder.
   * Known coagulopathy (e.g., hemophilia, von Willebrand disease) or platelet disorder relevant to aspirin use.
   * Platelet count <100,000/µL at screening.
   * Hemoglobin <8.0 g/dL at screening.
   * Current or anticipated need for full-dose anticoagulation (e.g., therapeutic low-molecular-weight heparin) or dual antiplatelet therapy during pregnancy.
3. Gastrointestinal / Hepatic / Renal

   * Active peptic ulcer disease, erosive esophagitis, or known upper GI lesion at significant risk for bleeding, not adequately treated.
   * History of recurrent peptic ulcer bleeding or perforation.
   * Documented cirrhosis or clinically significant chronic liver disease (e.g., Child-Pugh B or C).
   * Renal impairment, defined as Creatinine greater than 1.0 mg/dL, or currently on dialysis.
   * Known inflammatory bowel disease with recent moderate-severe flare (e.g., requiring steroids or hospitalization in the last 3 months).
4. Cardiovascular / Blood Pressure

   * Persistent severe hypertension at screening (e.g., ≥160/110 mmHg on repeated measurements) not adequately controlled on therapy.
   * Known significant structural heart disease or cardiomyopathy that, in the investigator's opinion, would increase risk with trial participation.
5. Pregnancy-Related / Obstetric

   * Multiple gestation (twins or higher-order).
   * Known major fetal structural anomaly or chromosomal abnormality at screening (if results already available).
   * Active preterm labor, preterm premature rupture of membranes (PPROM), or cervical dilation requiring emergent intervention at time of screening.
   * Placenta previa with active bleeding or high risk of bleeding where aspirin is contraindicated.
   * Planned elective termination of pregnancy.
   * Current or planned participation in an obstetric intervention that would make outcome attribution to the investigational regimen impossible (per investigator judgment).
6. Concomitant Medication Constraints (incl. CYP considerations)

   * Chronic daily use of aspirin >81 mg/day or other antiplatelet/NSAID therapy that cannot be discontinued or adjusted to comply with the protocol.
   * Current use of any PPI or H₂ blocker that cannot be safely discontinued or switched per protocol prior to randomization.
   * Concomitant use of medications with a very narrow therapeutic index that are strong CYP2C19 or CYP3A4 substrates and for which modest PK changes could pose significant risk (e.g., selected anticonvulsants, calcineurin inhibitors, or antiarrhythmics), where dose adjustment or close monitoring is not feasible.
   * Use of another investigational drug or device within 30 days prior to screening, or planned during the trial, that could affect maternal or fetal outcomes.
7. Other Medical Conditions

   * Any malignancy requiring active systemic therapy during pregnancy.
   * Uncontrolled autoimmune, rheumatologic, or hematologic disease that, in the opinion of the investigator, significantly increases risk with aspirin or PPI therapy.
   * Poorly controlled diabetes with significant end-organ complications (e.g., advanced nephropathy, proliferative retinopathy) where participation would add undue risk.
   * Any severe or unstable systemic illness (e.g., decompensated heart failure, severe pulmonary hypertension) that, in the investigator's judgment, makes trial participation unsafe.
8. Substance Use / Adherence

   * Active substance use disorder (alcohol or drugs) likely to interfere with adherence, follow-up, or maternal/fetal safety.
   * Any condition (including significant psychiatric illness or cognitive impairment) that, in the investigator's opinion, would compromise informed consent, adherence to study procedures, or reliable follow-up.
9. Study Conduct / Ethical Considerations

   * Concurrent participation in another interventional clinical trial impacting maternal-fetal outcomes.
   * Prior randomization in this trial during the current pregnancy.
   * Any other reason that, in the investigator's judgment, makes the participant unsuitable for the trial or at increased risk such that participation would not be in their best interest.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Eligibility to participate in this study is limited to pregnant individuals, regardless of gender identity. Participants must be able to become pregnant and be currently pregnant at the time of enrollment. Gender identity itself is not a criterion for inclusion or exclusion.
Enrollment: 670 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2030-09-30 (Estimated); Study Completion 2032-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with a diagnosis of Preterm Birth before 37+0 weeks of gestation | At or after 20+0 and before 37+0 weeks of gestation
  The primary endpoint is the incidence of preterm birth before 37+0 weeks of gestation, defined as delivery occurring at or after 20+0 and before 37+0 weeks of gestation, in biomarker-identified high-risk pregnant participants randomized to aspirin + lansoprazole versus standard of care.

SECONDARY OUTCOMES:
Incidence of preterm birth before 34+0 weeks of gestation. | Before 34+0 weeks of gestation.
  Incidence of preterm birth before 34+0 weeks of gestation.
Gestational age at delivery | At delivery
  Gestational age at delivery, analyzed as a continuous outcome (weeks).
Incidence of hypertensive disorders of pregnancy, including gestational hypertension, preeclampsia, and eclampsia. | At or after 20+0 and before 37+0 weeks of gestation
  Incidence of hypertensive disorders of pregnancy, including gestational hypertension, preeclampsia, and eclampsia.
Incidence of fetal growth restriction | At delivery.
  Incidence of fetal growth restriction, including:
  * Small-for-gestational-age (SGA; birthweight <10th percentile),
  * Low birthweight (<2500 g), and
  * Very low birthweight (<1500 g).

CONTACTS AND LOCATIONS:
Overall Officials: Brice Gaudillière, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: IPD Availability (Start Date): 6 months after publication of the primary results IPD Availability (End Date): 5 years after publication of the primary results
Access Criteria: Who can access:
  Qualified researchers (e.g., academic investigators or industry scientists) with a methodologically sound proposal and appropriate expertise, following review and approval by the study sponsor/investigator team.
  What they can access:
  De-identified, participant-level individual participant data (IPD) underlying the primary and secondary outcome results, along with supporting documentation such as the study protocol, statistical analysis plan, data dictionary/codebook, and analytic code as available.
  How access will be provided:
  Access will be granted upon submission of a written request and research proposal, completion of a data use agreement (DUA), and confirmation of IRB/ethics approval or exemption as applicable. Approved users will receive access via a secure data-sharing platform or encrypted file transfer, with use limited to the approved analyses and no attempts at re-identification permitted.
URL: https://gaudillierelab.stanford.edu/contact/